CLINICAL TRIAL: NCT06998966
Title: Quality Improvement Initiative Leveraging Electronic Healthcare Records to Reduce Inappropriate Proton Pump Inhibitors (PPI) Prescribing at UCLA.
Brief Title: Optimizing Proton Pump Inhibitors (PPI) Prescribing With EHR-Based Decision Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John N. Mafi, MD, MPH, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-25-0231; 1K76AG064392-01A1 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Prescribing Patterns, Physician; Physician's Practice Patterns; Drug Utilization Review
Keywords: Proton Pump Inhibitors; Quality Improvement; Healthcare Utilization; Clinical Decision Support; resource utilization

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): •Physicians use an unchanged prescribing workflow for Proton Pump Inhibitors (PPI) medications, with no changes to default dosage or duration.
- Algorithmic Defaulting (Indication-Based Default) (Experimental): The Electronic Health Record (EHR) automatically evaluates whether the patient at hand meets guideline criteria for long-term vs. short-term Proton Pump Inhibitors (PPI) use and it selects a default PPI prescription duration. (Providers can override the defaulted duration if they disagree with the automated assessment.) The order panel displays each PPI option below one of the following duration choices: For short-term PPI, this includes patients with conditions like Gastroesophageal reflux disease (GERD). For long-term PPI, this includes patients with conditions requiring extended therapy (e.g. Barrett's esophagus, chronic NSAID use)
  Interventions: Behavioral: Algorithmic Defaulting (Indication-Based Default)
- Active Physician Choice (Experimental): •The order panel displays each PPI option below one of the following duration choices: For short-term PPI, this includes patients with conditions like GERD. For long-term PPI, this includes patients with conditions requiring extended therapy (e.g. Barrett's esophagus, chronic NSAID use). The order panel removes the default selection, thus requiring providers to actively select a prescription duration for each patient, given the guideline education presented in the panel.
  Interventions: Behavioral: Active Physician Choice

INTERVENTIONS:
Behavioral: Algorithmic Defaulting (Indication-Based Default) — PPIs are frequently overprescribed, and the CareConnect default prescription setting of 90 days with three refills (360 pill days) exceed standard guidelines (in most cases, 60 pill days). It is unclear whether this is the most appropriate workflow. Given that deprescribing PPIs carries minimal risk for most patients, this initiative will assess whether modifying defaulted prescription lengths influences prescribing behavior while ensuring physicians retain full decision-making authority.
  Arms: Algorithmic Defaulting (Indication-Based Default)
Behavioral: Active Physician Choice — PPIs are frequently overprescribed, and the CareConnect default prescription setting of 90 days with three refills (360 pill days) exceed standard guidelines (in most cases, 60 pill days). It is unclear whether this is the most appropriate workflow. Given that deprescribing PPIs carries minimal risk for most patients, this initiative will assess whether requiring providers to actively select prescription lengths influences prescribing behavior while ensuring physicians retain full decision-making authority.
  Arms: Active Physician Choice

SUMMARY:
The proposed study is a quality improvement initiative designed to rigorously evaluate new variations of UCLA Health's proton pump inhibitor (PPI) order panels, building on internal quality improvement efforts to optimize prescribing workflows within the Electronic Health Record (EHR). PPIs are notoriously overprescribed, and the study team has identified that the CareConnect default prescription setting of 90 days with three refills (360 pill days) exceed standard guidelines (in most cases, 60 pill days). It is unclear whether this is the most appropriate workflow. Given that deprescribing PPIs carries minimal risk for most patients, this initiative will assess whether modifying defaulted prescription lengths influences prescribing behavior while ensuring physicians retain full decision-making authority.

This evaluation of PPI order panel variations is embedded within UCLA's existing EHR system, ensuring that changes are tested pragmatically within routine workflows. The study aims to determine whether small adjustments to the order panel can better align prescribing patterns with clinical best practices while maintaining physician autonomy.

ELIGIBILITY:
Inclusion Criteria:

* UCLA Health primary care physicians who have a clinical full-time equivalency of at least 25%.

Exclusion Criteria:

* Physicians with a clinical full-time equivalency of less than 25%

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Inappropriate Pill Days | 12 months
  The study will take place within the existing UCLA Health Electronic Health Record (EHR) infrastructure. Data will be automatically collected from the EHR, focusing on pill days in excess of guidelines. The trial team will validate an eMeasure of inappropriate prescriptions as the primary outcome.

SECONDARY OUTCOMES:
Prescription Discontinuations | 12 months
  The study will take place within the existing UCLA Health EHR infrastructure. Data will be automatically collected from the EHR, focusing on prescriptions that have been discontinued for 90 days or more.
Prescription Refills | 12 months
  The study will take place within the existing UCLA Health EHR infrastructure. Data will be automatically collected from the EHR, focusing on prescriptions that are refilled.
Overall Average Pill Days | 12 months
  The study will take place within the existing UCLA Health EHR infrastructure. Data will be automatically collected from the EHR, focusing on pill days overall.
GI Bleeding Hospitalization | 12 months
  Balancing measure to ensure reducing PPIs does not lead to harm.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No